CLINICAL TRIAL: NCT00543556
Title: MK0767 in Type 2 Diabetes (0767-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0767-012; 2007_640
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — MK0767

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0767

SUMMARY:
This is a clinical trial in patients with Type 2 Diabetes to test the safety of MK0767. This study will also see how effective MK0767 is in lowering markers of glucose metabolism and improving the lipid profile and non-HDL cholesterol when compared with placebo and pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus patients between the ages of 21 and 75 inclusive
* Patient is willing to discontinue current therapy for the duration of the study
* Patient is not a heavy drinker

Exclusion Criteria:

* Patient has a history of Type 1 diabetes and/or ketoacidosis
* Patient has severe diabetic retinopathy, or nephropathy, or neuropath
* Patient has has anti-hyperglycemic therapy including insulin, or rosiglitazone and pioglitazone or 2 or more oral agents in combination within 8 weeks prior to visit 1
* Patient has a history of, allergy to, intolerance or hypersensitive to troglitazone, rosiglitazone, or pioglitazone including history of elevated liver function test, jaundice, or hepatotoxicity associated with these treatments

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2001-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC